CLINICAL TRIAL: NCT04216212
Title: Is the Future of Gastroenterology Being Adequately Prepared to Prevent Work Related Injuries and Allow for a Long Healthy Career? Question Answered.
Brief Title: Gastroenterology & Work Related Injuries
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 058.GID.2018.D
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Gastroenterology & Work Related Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
2.2.1. Primary Outcome(s)

• Percentage of gastroenterology fellows who have received any formal training in the ergonomics of endoscopy and how to prevent long term work related injuries.

2.2.2. Secondary Outcome(s)

* How much formal training given in multiple choice format fellows received in the ergonomics of endoscopy and how to prevent work related injuries.
* Number of perceived work related injuries fellows sustained.
* Types of perceived work related injuries fellows sustained.
* If fellow perceived work related injuries whether they felt it negatively affected their ability to perform their duties as a gastroenterology fellow.

DETAILED DESCRIPTION:
This is a self-report survey utilizing a voluntary, non-probability sampling design. The survey instrument will be created in Google Survey© consisting of yes/no, multiple choice and free text response questions. This survey instrument questions have been developed empirically by the investigators.

It will be distributed to all gastroenterology fellowship coordinators through an email listserv maintained by programs nationwide for the purpose of communicating with their trainees. The email will include instructions to share the survey link (Appendix 2) with all first/second/third year as well as all advanced gastroenterology fellow s in their programs. The survey will be disseminated over a 2 week period. The fellowship coordinator will receive three separate emails. The first email (Appendix 2) will be on opening day of the survey requesting them to forward the link to their fellows. The second email (Appendix 3) will be sent on day 8 of the study period serving as a reminder to participate in the survey with link once again attached. The final email (Appendix 4) will be distributed on day 14 of the study period serving as a final reminder for fellows to complete the survey if they have not already and that the survey will close at midnight. The link will have both the informed consent form and the survey. Participants must press a key indicating agreement to get past the consent to the survey. The survey will take less than 2 minutes to complete electronically. This will be an anonymous survey and will be distributed via a secure online platform.

The results will be compiled using Google Survey© software. No personal identifying information will be included.

ELIGIBILITY:
Inclusion Criteria:

* Gastroenterology fellows enrolled in an accredited program in the United States
* First, second and third year as well as advanced gastroenterology fellows
* Able and willing to provide consent

Exclusion Criteria:

* Advanced gastroenterology fellows
* Staff gastroenterologists
* Unable or unwilling to provide consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: It will be distributed to all gastroenterology fellowship coordinators through an email listserv maintained by programs nationwide for the purpose of communicating with their trainees.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Training on ergonomics of endoscopy | 14 days
  • Percentage of gastroenterology fellows who have received any formal training in the ergonomics of endoscopy and how to prevent long term work related injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Craig, M.D., Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States